CLINICAL TRIAL: NCT07267052
Title: Acute Effects of Transcutaneous Electrical Nerve Stimulation at Acupoints on Nociceptive Transmission: A Mechanism Study Using Pain-Related Evoked Potentials
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: China Medical University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CMUH114-REC3-149
Record Dates: First submitted 2025-11-25; First posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Pain Management
Keywords: Somatosensory Evoked Potentials; Transcutaneous Electrical Nerve Stimulation; Pain-Related Evoked Potentials; Zhongzhu; Hegu
MeSH Terms: conditions — Agnosia | interventions — Transcutaneous Electric Nerve Stimulation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- TENS Group (Experimental): Acupoint TENS Intervention (TENS Group) Participants in this group received low-frequency transcutaneous electrical nerve stimulation (TENS) applied to clinically recognized analgesic acupoints, Zhongzhu (SJ3) and Hegu (LI4). Each participant completed two intervention sessions in a randomized order, with at least 48 hours between sessions. During each session, participants first underwent a baseline assessment of pain-related evoked potentials (PREPs), followed by a 20-minute TENS application delivered through surface electrodes placed directly over the target acupoint. The stimulation parameters included low frequency and low-intensity currents adjusted to a comfortable but perceptible level. Immediately after the stimulation period, participants received a follow-up PREP assessment to evaluate changes in nociceptive cortical processing. Subjective pain responses and any discomfort or adverse reactions were recorded throughout the procedure. The entire protocol was designed to deter
  Interventions: Device: transcutaneous electrical nerve stimulation (TENS); Device: EEG machine

INTERVENTIONS:
Device: transcutaneous electrical nerve stimulation (TENS) — TENS was applied to the acupoints Zhongzhu (SJ3) and Hegu (LI4) using surface electrodes. Low-frequency electrical currents were delivered at an intensity that was comfortable but perceptible, without causing muscle contraction. Each session lasted 20 minutes, during which participants remained seated and relaxed, and electrode placement and stimulation parameters were monitored for safety and consistency.
Device: EEG machine — EEG signals were recorded using the Neuro-MEP4 system. The device captures cortical electrical activity with high temporal resolution and is suitable for measuring pain-related evoked potentials (PREPs). Standard electrode placement and recording protocols were followed, and signal quality was checked before each session to ensure reliable data collection.

SUMMARY:
The goal of this clinical trial is to learn if transcutaneous electrical nerve stimulation (TENS) applied to acupoints can modulate pain transmission and cortical processing in healthy adult volunteers. The main questions it aims to answer are:

* Does TENS at Zhongzhu (SJ3) and Hegu (LI4) change pain-related evoked potentials (PREPs)?
* Does acupoint electrical stimulation alter nociceptive pathways reflected by PREP waveform modulation?

Researchers will compare PREPs recorded before and after TENS at the two acupoints to see if TENS produces measurable effects on cortical nociceptive responses.

Participants will receive low-frequency TENS applied to Zhongzhu (SJ3) and Hegu (LI4), and undergo PREP assessments before and after the intervention to measure cortical responses to standardized noxious stimuli.

DETAILED DESCRIPTION:
This study aims to investigate the modulatory effects of transcutaneous electrical nerve stimulation (TENS) applied to acupuncture points on pain transmission and cortical processing in healthy adults. Pain-related evoked potentials (PREPs) will be used as the primary neurophysiological measure to examine changes before and after TENS applied to two clinically recognized analgesic acupoints, Zhongzhu (SJ3) and Hegu (LI4). A within-subject design will be adopted, and participants aged 18 years or older will undergo two experimental sessions in randomized order. Each session will include baseline PREP assessment, a 20-minute low-frequency TENS intervention at the assigned acupoint, and a follow-up PREP measurement. PREP waveform characteristics, including N2 and P2 amplitudes and latencies, will be analyzed to determine whether acupoint stimulation alters nociceptive transmission. Subjective pain reports and adverse responses will also be collected to assess tolerability. The findings of this research are expected to provide insight into the neurophysiological basis of acupuncture analgesia and contribute to the development of more refined acupoint-based electrical therapies.

ELIGIBILITY:
Inclusion Criteria:

* Participants will be healthy adults aged 20 years or older. All participants must meet the inclusion criteria, including the absence of chronic medical conditions, no history of drug allergies or skin disorders, and no current use of medications that could affect study outcomes. To ensure the reliability of the results, participants are required to maintain a regular daily routine and have no history of substance or medication abuse.

Exclusion Criteria:

* Participants with a history of malignant tumors, hand disorders, implanted cardiac pacemakers, pregnancy, epilepsy, or any other condition that may interfere with the study procedures will be excluded from the study.

Min Age: 20 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 35 (Estimated)
Dates: Start 2025-11-25 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Pain-Related Evoked Potentials (PREPs) | Participants were assessed at time points: prior to the intervention (baseline), immediately after TENS application
  PREPs were recorded using the Neuro-MEP4 EEG system. Participants were seated comfortably in a quiet room and instructed to remain relaxed during the recordings. Surface electrodes were placed according to standard PREP protocols to capture cortical responses to standardized noxious electrical stimuli applied to the forearm. For each trial, multiple stimuli were delivered, and the resulting N2 and P2 components were averaged to improve signal reliability. The primary outcome measures included the peak amplitudes and latencies of the N2 and P2 waves, which reflect cortical processing of nociceptive input.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Physical Therapy of China Medical University, Taichung, Beitun, Taiwan, Taiwan